CLINICAL TRIAL: NCT03261271
Title: Weight Management Aimed to Reduce Risk and Improve Outcomes From Radical Prostatectomy
Acronym: WARRIOR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Collaborators: American Cancer Society, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: STUDY00141060; RSG-17-050-01-NEC (Other Grant/Funding Number: American Cancer Society)
Record Dates: First submitted 2017-08-22; First posted 2017-08-24 (Actual); Results first posted 2025-02-26 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2025-04

CONDITIONS: Obesity; Prostate Cancer
MeSH Terms: conditions — Obesity; Prostatic Neoplasms | interventions — Weight Reduction Programs

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Weight Loss and Weight Maintenance (Experimental): Participants will take part in a weight loss program for at least 4 weeks (and up to 16 weeks) before their prostatectomy, and a weight maintenance program for 6 months after their surgery.
  Interventions: Behavioral: Weight Loss Program; Behavioral: Weight Maintenance Program
- Control (Active Comparator): Participants will receive a standardized educational flyer about a healthy diet and exercise.
  Interventions: Behavioral: Standardized educational flyer

INTERVENTIONS:
Behavioral: Weight Loss Program — Program involves one-on-one coaching, diet meal plan, and physical activity plan.
  Arms: Weight Loss and Weight Maintenance
Behavioral: Standardized educational flyer — The American Institute for Cancer Research handout "Nutrition and the Cancer Survivor" will be provided to participants.
  Arms: Control
Behavioral: Weight Maintenance Program — Post-surgery program involves group support sessions, phone check-ins, and diet and exercise monitoring.
  Arms: Weight Loss and Weight Maintenance

SUMMARY:
The purpose of this study is to test how a weight management program affects substances in the blood called biomarkers that can show the presence or severity of cancer, compared to a standardized diet and exercise educational flyer.

ELIGIBILITY:
Inclusion Criteria:

* Men newly diagnosed with PCa who are scheduled for radical prostatectomy (RP) (T1 or T2)
* Body Mass Index (BMI) 25-45 kg/m2
* Has internet access

Exclusion Criteria:

* History of 5 alpha reductase inhibitors prior 3 months
* History of radiation therapy for cancer treatment
* Taking active cancer treatment
* Undergoing salvage therapy
* Castration-resistant PCa
* Evidence of metastasis
* Evidence of biochemical recurrence
* High risk medical condition (e.g. kidney disease, uncontrolled diabetes, etc.)

Min Age: 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 40 (Actual)
Dates: Start 2017-11-02 (Actual); Primary Completion 2023-11-28 (Actual); Study Completion 2025-03-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jill Hamilton-Reeves, PhD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participant enrollment took place from November 2017 to August 2020 at The University of Kansas Health System. Participants were recruited from the Department of Urology medical clinic.
Pre-assignment Details: Upon enrollment, participants were randomized to either the intervention or active control arms.
Period: Overall Study
Arm/Group | Weight Loss and Weight Maintenance | Control
Started | 20 | 20
Completed | 19 | 19
Not Completed | 1 | 1
Not completed — Treatment changed after surgery. Participants were removed from the study. | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Weight Loss and Weight Maintenance | Control | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.25 (5.86) | 60.80 (5.66) | 60.03 (5.74)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 20 | 20 | 40
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 20 | 19 | 39
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 2 | 3
  White | 18 | 18 | 36
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 20 | 20 | 40
Highest Education Level [Count of Participants; unit: Participants]
  High School/GED | 2 | 3 | 5
  Some College/Associate's | 10 | 7 | 17
  Bachelor's | 4 | 7 | 11
  Master's | 4 | 2 | 6
  Doctoral | 0 | 0 | 0
  Not reported | 0 | 1 | 1
Rural-Urban Commuting Area (RUCA) Codes [Count of Participants; unit: Participants] — RUCA codes are a census tract-based classification that uses standard census measures of population density, levels of urbanization and daily commuting patterns. Codes range from 1 (highly urban) to 10 (highly rural).
  Participants
    RUCA Code 1 | 12 | 13 | 25
    RUCA Code 2 | 7 | 2 | 9
    RUCA Code 4 | 0 | 1 | 1
    RUCA Code 7 | 1 | 2 | 3
    RUCA Code 10 | 0 | 2 | 2
Smoking Status [Count of Participants; unit: Participants]
  Current Smoker | 2 | 1 | 3
  Former Smoker | 8 | 10 | 18
  Never Smoked | 10 | 9 | 19
Preoperative Erectile Dysfunction [Count of Participants; unit: Participants] | 9 | 10 | 19
Prostate Specific Antigen (PSA) [Mean (Standard Deviation); unit: ng/mL] | 7.96 (5.76) | 8.31 (6.09) | 8.14 (5.85)
Gleason score [Mean (Standard Deviation); unit: units on a scale] — A Gleason score is a grading system used to describe prostate cancer and determine its aggressiveness. Gleason scores range from 2-10. Pathologists rarely assign scores 2-5. Gleason scores assigned will range from 6 to 10, with 6 being low grade, 7 intermediate grade, and a score of 8 to 10 is high grade cancer.
  units on a scale | 7.05 (0.76) | 7.05 (0.22) | 7.05 (0.55)
Weight [Mean (Standard Deviation); unit: kg] | 106.94 (17.15) | 101.54 (10.42) | 104.24 (14.27)
Height [Mean (Standard Deviation); unit: cm] | 177.38 (6.60) | 176.55 (4.45) | 176.96 (5.57)
BMI [Mean (Standard Deviation); unit: kg/m2] | 33.95 (4.90) | 32.59 (3.29) | 33.27 (4.18)

OUTCOME MEASURES:

1. Primary Outcome: Impact of Weight Loss Before and Weight Maintenance After Prostate Cancer (PCa) Surgery on Immunosuppressive Factors
Description: Impact will be measured by changes in specific blood immune biomarker monocytic myeloid-derived suppressor cells (mMDSCs). The absolute number of cell counts were calculated using the lymphocyte count abstracted from the complete blood count with differential.
Time Frame: Change from Baseline to Month 6
Population: Intent to Treat Population (all participants assigned to Weight Loss and Weight Maintenance or Control).
Measure: Mean (Standard Deviation); unit: count of cells
Arm/Group | Weight Loss and Weight Maintenance | Control
Number analyzed (Participants) | 20 | 20
count of cells
  Baseline mMDSC count: number analyzed (Participants) | 20 | 19
  Baseline mMDSC count | 19.29 (26.72) | 17.37 (18.96)
  1 week prior to surgery mMDSC count: number analyzed (Participants) | 19 | 20
  1 week prior to surgery mMDSC count | 17.68 (21.14) | 12.76 (15.64)
  6 months after surgery mMDSC count: number analyzed (Participants) | 17 | 17
  6 months after surgery mMDSC count | 40.52 (44.87) | 32.91 (36.38)
Statistical Analysis 1: Comparison: Weight Loss and Weight Maintenance vs Control; Test type: Superiority; p = 0.6489, Mixed Models Analysis — P value less than 0.05 was considered statistically significant

2. Secondary Outcome: Impact of Weight Loss Before and Weight Maintenance After PCa Surgery on Inflammation Factors
Description: Impact will be measured by changes in specific blood biomarker leptin/adiponectin ratio.
Time Frame: Change from Baseline to Month 6
Population: Intent to Treat Population (all participants assigned to Weight Loss and Weight Maintenance or Control).
Measure: Mean (Standard Deviation); unit: leptin/adiponectin ratio
Arm/Group | Weight Loss and Weight Maintenance | Control
Number analyzed (Participants) | 20 | 20
leptin/adiponectin ratio
  Baseline leptin/adiponectin ratio | 0.28 (0.29) | 0.28 (0.27)
  1 week prior to surgery leptin/adiponectin ratio: number analyzed (Participants) | 20 | 19
  1 week prior to surgery leptin/adiponectin ratio | 0.16 (0.21) | 0.29 (0.22)
  6 months after surgery leptin/adiponectin ratio: number analyzed (Participants) | 18 | 17
  6 months after surgery leptin/adiponectin ratio | 0.11 (0.14) | 0.25 (0.32)
Statistical Analysis 1: Comparison: Weight Loss and Weight Maintenance vs Control; Test type: Superiority; p = 0.0323, Mixed Models Analysis

3. Secondary Outcome: Change in Weight
Description: Body weight will be measured at participant study visits.
Time Frame: Change from Baseline to Month 6
Population: Intent to Treat Population (all participants assigned to Weight Loss and Weight Maintenance or Control).
Measure: Mean (Standard Deviation); unit: weight in kilograms
Arm/Group | Weight Loss and Weight Maintenance | Control
Number analyzed (Participants) | 20 | 20
weight in kilograms
  Baseline body weight (kg) | 106.9 (17.2) | 101.5 (10.4)
  1 week prior to surgery body weight (kg) | 101.1 (16.5) | 100.6 (11.1)
  6 months after surgery body weight (kg): number analyzed (Participants) | 19 | 18
  6 months after surgery body weight (kg) | 95.8 (17.5) | 99.8 (11.1)
Statistical Analysis 1: Comparison: Weight Loss and Weight Maintenance vs Control; Test type: Superiority; p < 0.0001, Mixed Models Analysis

4. Secondary Outcome: Change in Body Composition
Description: Body composition will be measured using a Dual Energy X-Ray Absorptiometry (iDXA). Change in percent body fat will be analyzed between groups from baseline to study end.
Time Frame: Change from Baseline to Study End
Population: Intent to Treat Population (all participants assigned to Weight Loss and Weight Maintenance or Control).
Measure: Mean (Standard Deviation); unit: percentage of body fat
Arm/Group | Weight Loss and Weight Maintenance | Control
Number analyzed (Participants) | 20 | 20
percentage of body fat
  Baseline body fat % | 39.2 (4.9) | 37.6 (4.3)
  1 week prior to surgery body fat % | 37.1 (5.4) | 37.4 (4.8)
  6 months after surgery body fat %: number analyzed (Participants) | 18 | 17
  6 months after surgery body fat % | 34.0 (7.6) | 36.7 (4.2)
Statistical Analysis 1: Comparison: Weight Loss and Weight Maintenance vs Control; Test type: Superiority; p < 0.0001, Mixed Models Analysis

5. Secondary Outcome: Change in Quality of Life
Description: Quality of Life will be measured using the Expanded PCa Index Composite (EPIC) Instrument-26. There are a total of 26 items on the survey. Scores range from 0 to 100. The higher the score, the higher the quality of life.
Time Frame: Change from Baseline to Month 6
Population: Intent to Treat Population (all participants assigned to Weight Loss and Weight Maintenance or Control).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Weight Loss and Weight Maintenance | Control
Number analyzed (Participants) | 20 | 20
units on a scale
  General Health Quality of Life at Baseline | 47.8 (7.0) | 48.0 (7.8)
  General Health Quality of Life at Pre-Surgery | 52.5 (6.0) | 48.6 (8.5)
  General Health Quality of Life at Study End | 52.0 (8.6) | 47.7 (8.9)
Statistical Analysis 1: Comparison: Weight Loss and Weight Maintenance vs Control; Difference between groups from Baseline to Study End; Test type: Superiority; p = 0.09, Mixed Models Analysis
Statistical Analysis 2: Comparison: Weight Loss and Weight Maintenance vs Control; Difference between groups from baseline to pre-surgery; Test type: Superiority; p = 0.04, Mixed Models Analysis

ADVERSE EVENTS:
Time Frame: 4-16 weeks prior to surgery and 6 months after surgery. At most, 10 months.
Description: Adverse Events were not assessed for the control group since they did not follow the study intervention. The control group received educational materials and followed standard of care.
Arm/Group | Weight Loss and Weight Maintenance
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 7/20
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Weight Loss and Weight Maintenance (N=20)
Constipation (Gastrointestinal disorders) | 2 (2)
Bloating (Gastrointestinal disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (2)
Muscle pain or strain (Musculoskeletal and connective tissue disorders) | 4 (4)

LIMITATIONS AND CAVEATS:
This randomized controlled trial could not be blinded to participants due to the nature of the intervention.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-03-23): https://cdn.clinicaltrials.gov/large-docs/71/NCT03261271/Prot_SAP_000.pdf
  • Informed Consent Form (2019-09-03): https://cdn.clinicaltrials.gov/large-docs/71/NCT03261271/ICF_001.pdf